CLINICAL TRIAL: NCT04330885
Title: PRE Surgery reHABilitation for Patients Suffering From Spinal Stenosis
Brief Title: PRE Surgery reHABilitation for Spinal Stenosis
Acronym: PreShab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Rasmussen Barr, Associated professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLS-683231
Record Dates: First submitted 2019-12-31; First posted 2020-04-02 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain; Rehabilitation; Physiotherapy
Keywords: prehabilitation; spinal stenosis; physiotherapy
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with two treatment arms; one with care as usual and the intervention group with prehab before surgery. This is a feasibility study to determine how many subjects who need to be included to be able to a obtain an estimate of variance in an outcome when an important difference between groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator does not take part in data collection. All data collected via web based surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehab group (Experimental): The patients in the PREHAB group will meet with a PT for 6 weeks pre surgery. The PT will coach the patient in 1:1 visits with a graded activity program with the purpose to affect fear of movement and raising level of self-efficacy with physical activity. The intervention comprises; cycling on a stationary cycle. Instructions of exercises that strengthen the deep and the superficial abdominal muscles and the back muscles. Information to contract the abdominal muscles in posturally loaded position to support their back. Information on flexion exercises of their lumbar spine and to keep the back in a flexed position when standing and walking (as opposed to extension). Recommendation to use "Nordic walk (stavar)" for outdoor walking
  Interventions: Other: Supervised abdominal exercises and stationary biking
- Care as usual (No Intervention): Control group will be treated with care as usual meaning information from a PT two weeks prior to the surgery with information on the surgery and to stay active. Both groups will be given information on to stay active and home exercises following the surgery.

INTERVENTIONS:
Other: Supervised abdominal exercises and stationary biking — Explain pain to the patients in order to minimize fear of movement
  Other Names: Explain pain
  Arms: Prehab group

SUMMARY:
Lumbar spinal stenosis is a spinal disorder that affects mainly people over the age of 60. LSS is the most common reason to perform spinal surgery for people aged >65 years and have been shown to be superior to conservative treatment. Hitherto, studies on lumbar spinal stenosis are sparse with only 3 trials including approximately 300 patients. There is also a paucity in studies investigating if people with lumbar spinal stenosis improve their outcome following surgery undergoing a pre-surgery rehabilitation programme including physical fitness exercises, abdominal and back muscle strengthening and a core control approach.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a spinal disorder that affects mainly people over the age of 60. This age group with neurogenic claudication is expected to rise dramatically over the next 20 years when an estimated 23-25 % of the population will be > 60 years. Lumbar spinal stenosis is the most common reason to perform spinal surgery for people aged >65 years and have been shown to be superior to conservative treatment. Conservative treatment post-operatively have recently been described in a Cochrane review to be of importance. Hitherto, studies on lumbar spinal stenosisare sparse with only 3 trials including approximately 300 patients. There is also a paucity in studies investigating if people with lumbar spinal stenosis improve their outcome following surgery undergoing a pre-surgery rehabilitation programme including physical fitness exercises, abdominal and back muscle strengthening and a core control approach.

Aim: The aim of the current study was to evaluate a pre-surgery rehabilitation intervention for patients diagnosed with lumbar spinal stenosis found eligible for a decompression surgery. A further aim was to conduct a qualitative study to explore the experience of symptoms in relation to all-day-living and quality of life among those who have undergone a decompression surgery for lumbar spinal stenosis.

Methods: Patients consecutively seeking or referred for orthopaedic surgery at Spine Clinic in Stockholm will, if found eligible and given their informed consent be randomized into two separate groups following a consultant visit to an orthopaedic surgeon; 1) A pre-habilitation program of 8 weeks before decompression surgery 2) Care as usual, that is information from physiotherapists 2 weeks before surgery and the advice to stay active. Those eligible for decompression surgery are patients aged 50-75 with pseudo-claudication in one or both legs and back pain (VAS>30), magnetic resonance camera with 1-2 adjacent stenotic segments (L3-S1) (area ≤75mm2), duration of symptoms >6 months.

Both written and oral information of the study will be given and the patients will give their written consent. An independent physiotherapist blinded to patient assignment will sequentially number the envelopes containing intervention assignments according to a computer-generated randomization. Opaque and sealed envelopes will be opened in front of the participants at the end of the initial assessment visit. The main applicant will be responsible for data collection, to set up the program and educate included physiotherapists, to be responsible for analyses of data and for ethical application.

For the secondary aim a strategic sample of patients from both groups following the surgery will be included to conduct semi-structured deep interviews to explore their experience of facilitators and barriers to every day life both before and after the surgery. The interviews will take place 3 months following the surgery. The collected data will be analysed according a content analysis with categories, sub categories and themes.

ELIGIBILITY:
Inclusion Criteria:

* Spinal stenosis
* Eligible for decompression surgery
* aged 50-75 years
* pseudo-claudication in one or both legs
* back pain (VAS>30),
* MRI with 1-2 adjacent stenotic segments (L3-S1) (area ≤75mm2),
* duration of symptoms >6 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Change of Pain level: Numeric pain rating scale 0-11 | 6 weeks pre-surgery, pre-surgery, 3 and 12 months after surgery
  Numeric pain rating scale 0-10, higher value means more pain
Change of Disability level | 6 weeks pre-surgery, pre surgery, 3 and 12 months after surgery
  Oswestry Disability Index 0-100, higher value means more functional limitations

SECONDARY OUTCOMES:
Change of Fear of movement | 6 weeks pre-surgery, pre-surgery, 3 and 12 months after surgery
  Fear Avoidance Belief Questionnaire physical activity 0-25, higher score indiactes higher fear
Change of Self efficacy: Self efficacy scale 0-64 | 6 weeks pre-surgery, pre-surgery, 3 and 12 months after surgery
  Self efficacy scale for physical activity in low-back pain,higher value indicates a better self-efficacy
Change of General Health higher value means better health | 6 weeks before surgery, pre surgery, 3 and 12 months after surgery. HIgher values menas better health
  EuroQol-5 Dimensions Index (EQ5D), 3-point adjectival scale

OTHER OUTCOMES:
Global Change on a Likert Scale 5 point scale from not changed at all to changed fully | 12 months after surgery
  Global recovery, Question to value the overall change of symtoms, measured with Likert scale of 5 steps. HIgher value means better global recovery
Change of 6 minutes walk test Longer distance means better outcome. | 6 weeks pre-surgery, pre -surgery, 3 and 12 months after surgery
  Walk test - , assessed distance managed on 6 minutes, self chosen pace

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rasmussen Barr, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Ryggkirurgiskt Centrum, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No